CLINICAL TRIAL: NCT06514521
Title: A Post Marketing Surveillance on PluvictoTM (Lutetium(177Lu) Vipivotide Tetraxetan) in South Korea; An Open-label, Non-interventional, Primary Data Collection, Multi-center, Non-comparative, Non-randomized Observational Study to Assess Safety and Effectiveness of Pluvicto in Real World Setting
Brief Title: Post Marketing Study on Pluvicto in Korea
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAAA617A1KR01
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Metastatic castration-resistant prostate cancer; mCRPC; PMS; RMP; Pluvicto; Korea
MeSH Terms: interventions — Pluvicto

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lutetium vipivotide tetraxetan: Patients prescribed with Lutetium vipivotide tetraxetan in real world practice
  Interventions: Other: Lutetium vipivotide tetraxetan

INTERVENTIONS:
Other: Lutetium vipivotide tetraxetan — This is an observational study. There is no treatment allocation. The decision to initiate Lutetium vipivotide tetraxetan will be based solely on clinical judgement.
  Other Names: Pluvicto

SUMMARY:
Post marketing study on Pluvicto in Korea

DETAILED DESCRIPTION:
This is open-label, multi-center, non-comparative, non-interventional observational study to assess safety and effectiveness of Pluvicto in patients with mCRPC in the real-world setting in South Korea.

ELIGIBILITY:
Inclusion criteria

Study participants eligible for inclusion in this study must meet all of the following criteria:

1. Male adult patient age ≥ 18
2. Subject who are being treated with Pluvicto or whose treatment plan is finalized and scheduled to be administered at the time of consent by physician in accordance with the approved indication in South Korea
3. Subject who provided the written informed consent prior to the study enrollment

Exclusion criteria

Study participants meeting any of the following criteria are not eligible for inclusion in this study:

1. Subject whose medical record is not accessible
2. Subject who is not willing to provide the informed consent

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been using or going to receive Pluvicto per clinical judgment under routine medical practice are eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 278 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Serious Adverse Events, unexpected Adverse Events, Adverse Drug Reactions, Serious Adverse Drug Reactions and unexpected Adverse Drug Reactions | Until 30 days after the last dose of Pluvicto, up to 33 months
  The safety assessment will consist of occurrence status of all adverse events (AEs)/adverse drug reactions (ADRs), serious AEs (SAEs)/serious ADRs and unexpected AEs/unexpected ADRs.
  Safety data will be collected from all subjects over the study period. Subjects will be followed up for AEs until 30 days after the last dose of Pluvicto.

SECONDARY OUTCOMES:
Objective response rate (ORR) as assessed by investigator | 4th±1 week from the last dose
  Clinical assessment on disease status by investigator will be collected to assess objective response rate (ORR). If results are not available at study schedule, the nearest and available data will be collected. In case of subject follow up loss or discontinuation for any reason, ORR will be assessed based on the data collected at the date of the last contact of the subject.
Radiographic progression-free survival (rPFS) | Up to 33 months
  rPFS, defined as the time from study assignment to the date when the first sign of disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- South Korea (4):
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Seoul

IPD SHARING:
Plan to Share IPD: No